CLINICAL TRIAL: NCT07015294
Title: Effects of a Fruit- and Vegetable-Based Diet With Chaya Supplementation on Genomic Instability Indices and Biochemical Parameters in Breast Cancer Patients Undergoing Neoadjuvant Treatment
Brief Title: Effect of a Fruit- and Chaya-Based Diet on Genomic Instability and Biochemical Markers in Women With Breast Cancer Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anahuac Mayab University (Other)
Responsible Party: Principal Investigator, Elda Leonor Pacheco Pantoja, Senior Researcher, Anahuac Mayab University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 092024
Record Dates: First submitted 2025-05-26; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Cnidoscolus chayamans; Genomic instability
MeSH Terms: conditions — Breast Neoplasms; Genomic Instability | interventions — Fruit

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet rich in fruits and chaya infusion (Experimental): Participants followed a diet emphasizing increased fruit consumption and daily intake of chaya infusion (prepared from Cnidoscolus chayamansa leaves), known for its potential antioxidant properties. The diet was maintained throughout neoadjuvant chemotherapy cycles
  Interventions: Dietary Supplement: Fruits and chaya infusion
- Conventional diet (Active Comparator): Participants continued their usual dietary habits, with no specific modifications, throughout the course of neoadjuvant chemotherapy
  Interventions: Dietary Supplement: Conventional diet

INTERVENTIONS:
Dietary Supplement: Fruits and chaya infusion — Increased fruit consumption and daily intake of chaya infusion (prepared from Cnidoscolus chayamansa leaves),
  Arms: Diet rich in fruits and chaya infusion
Dietary Supplement: Conventional diet — Usual dietary habits, with no specific modifications
  Arms: Conventional diet

SUMMARY:
This exploratory, non-randomized clinical study aims to evaluate the potential impact of a diet enriched with fruits and chaya (Cnidoscolus aconitifolius) infusion on genomic instability and selected biochemical parameters in women with breast cancer undergoing neoadjuvant chemotherapy (NAC). Participants are assigned to either a control group receiving a conventional diet or an experimental group receiving the modified diet. Blood samples are collected at three time points during chemotherapy: prior to the first session, after the second cycle, and after the third cycle. The study involves the analysis of genomic instability using the comet assay, along with standard hematological and biochemical testing.

The study was reviewed and approved by the Research Ethics Committee of the Graduate and Research Unit of the Faculty of Medicine at the Universidad Autónoma de Yucatán. It is being conducted between August 2022 and September 2024.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 20-65 years
* Histologically confirmed breast cancer diagnosis
* Scheduled to undergo neoadjuvant chemotherapy
* Ability to consume chaya infusion and fruits as part of diet
* Provided informed consent

Exclusion Criteria:

* Diabetes mellitus or other uncontrolled metabolic diseases
* Severe hepatic or renal insufficiency prior to NAC
* Allergy or intolerance to any component of the experimental diet
* Participation in other clinical trials during the study period

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants
Enrollment: 13 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Genomic instability index (Comet assay) | Baseline (prior to first NAC cycle), at the end of Cycle 2 (approximately Day 42), and at the end of Cycle 3 (approximately Day 63); each NAC cycle is 21 days in duration.
  Measurement of DNA damage in peripheral blood leukocytes using the Comet assay, reported as tail length and tail moment

SECONDARY OUTCOMES:
Serum creatinine levels | Baseline (prior to first NAC cycle), at the end of Cycle 2 (approximately Day 42), and at the end of Cycle 3 (approximately Day 63); each NAC cycle is 21 days in duration.
  To assess kidney function during NAC under different dietary conditions.
Serum aspartate aminotransferase levels | Baseline (prior to first NAC cycle), at the end of Cycle 2 (approximately Day 42), and at the end of Cycle 3 (approximately Day 63); each NAC cycle is 21 days in duration.
  To evaluate hepatic enzyme fluctuations associated with diet and chemotherapy
Blood glucose levels | Baseline (prior to first NAC cycle), at the end of Cycle 2 (approximately Day 42), and at the end of Cycle 3 (approximately Day 63); each NAC cycle is 21 days in duration.
  To evaluate glycemia fluctuations associated with diet and chemotherapy
Hemoglobin | Baseline (prior to first NAC cycle), at the end of Cycle 2 (approximately Day 42), and at the end of Cycle 3 (approximately Day 63); each NAC cycle is 21 days in duration.
  To assess hematologic stability during the intervention period.
Serum alanine aminotransferase levels | Baseline (prior to first NAC cycle), at the end of Cycle 2 (approximately Day 42), and at the end of Cycle 3 (approximately Day 63); each NAC cycle is 21 days in duration.
  To evaluate hepatic enzyme fluctuations associated with diet and chemotherapy
Platelet counts | Baseline (prior to first NAC cycle), at the end of Cycle 2 (approximately Day 42), and at the end of Cycle 3 (approximately Day 63); each NAC cycle is 21 days in duration.
  To assess hemostasis stability during the intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Anahuac Mayab, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in this study (including text, tables, figures, and appendices) will be made available to researchers upon reasonable request.
Supporting Information: SAP